CLINICAL TRIAL: NCT06538064
Title: A Global Real-World Study to Assess HyQvia Use and Outcomes in Patients With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) Switching to HyQvia
Brief Title: A Study of HyQvia in Adults With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) in Routine Clinical Care
Acronym: HYbISCUE
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-771-5008; 2024-512690-26-00 (EU CTIS Number: EUCTR Number)
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: New Users of HyQvia: Participants with CIDP who intend to switch to HyQvia within 6 weeks after enrollment will be interviewed and data from medical records will be reviewed for 12 months.
  Interventions: Other: No Intervention
- Cohort B: Current Users of HyQvia: Participants with CIDP who switched to HyQvia within 6 weeks prior to enrollment will be interviewed and data from medical records will be reviewed for 12 months.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The main aims of this study are to understand why adults with Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) chose a certain treatment, why they changed to HyQvia from another therapy, how satisfied they are with HyQvia and their previous treatment, how their work productivity and activity is impacted and learn about their CIDP signs and symptoms. Other aims are to collect information on any medical problems or side effects during the treatment with HyQvia, learn how effective treatment of CIDP with HyQvia is and understand details on the use of HyQvia in standard clinical routine as well on the need for healthcare intervention (such as emergency room visits or hospital visits or stays).

During the study, data will be collected from medical records already available, interviews with participants at study start and study completion and via questionnaires completed by participants.

Participants will be treated as per the doctor's or the clinic's routine.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or older.
* Investigator-confirmed documented diagnosis of CIDP of any type (e.g., typical, multifocal, focal, motor, sensory, or distal) according to the revised European Academy of Neurology and Peripheral Nerve Society (EAN/PNS) 2021 guidelines on the diagnosis and treatment of CIDP.
* Participants must currently have a stable disease course (as per physician judgment) for at least 12 weeks.
* Is considered a new user or current user of HyQvia-

  * New users (Cohort A) are participants on a CIDP treatment as of the date of enrollment, who intend to switch to HyQvia within 6 weeks after enrollment.
  * Current users (Cohort B) are participants on HyQvia as of the date of enrollment, who switched to HyQvia within the 6 weeks preceding the date of enrollment (the 6-week window may be extended depending on the recruitment progress).
* Has provided written informed consent (for the main study).
* Participant is willing to comply with the protocol requirement of non-standard of care (non-SOC) assessments (e.g., adjusted inflammatory neuropathy cause and treatment (INCAT) assessment).
* Participants must be able to communicate fluently in their local language (if they participate in the optional qualitative participant interview [sub-study].

Exclusion Criteria:

* Had any HyQvia use, defined as

  * any record of HyQvia use prior to enrollment for new users of HyQvia (Cohort A), and
  * any record of HyQvia use more than 6 weeks preceding the enrollment date (the 6-week window may be extended depending on the recruitment progress) for current users of HyQvia (Cohort B).
* Without any prior treatment for CIDP.
* Pregnant or breastfeeding.
* Participants with known hypersensitivity to any component of HyQvia.
* Has participated in an interventional clinical study within 30 days prior to enrollment or was scheduled to participate in an interventional clinical study during this study.
* Has had major surgery within 12 weeks prior to enrollment, or has surgery planned during the time the participant is expected to participate in the study. Note: Participants with planned surgical procedures to be conducted under local anesthesia may participate. Kyphoplasty or vertebroplasty are not considered major surgeries.
* Received induction treatment for CIDP during the past 12 weeks.
* Participant is identified by the investigator as being unable or unwilling to cooperate with the study procedures.
* (Cohort A) only: Participants who do not initiate HyQvia treatment within 6 weeks after enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is participants with a confirmed clinical diagnosis of CIDP, who are in the process of switching from any prior CIDP therapy to HyQvia for maintenance treatment of CIDP. The participants population will be comprised of both new users (Cohort A) and current users (Cohort B) of HyQvia.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-08-17 (Estimated); Study Completion 2027-08-17 (Estimated)

PRIMARY OUTCOMES:
Treatment Preference for CIDP Therapy as Measured by Novel Treatment Preference Questionnaires | Baseline up to 12 months (HyQvia or study discontinuation)
  The novel treatment preference questionnaires measure participant's treatment preferences for switching to HyQvia from other subcutaneous immunoglobulin/intravenous immunoglobulin (SCIG/IVIG) treatments for CIDP. It includes overall preference for switching from prior therapy to HyQvia, reason for switching from prior therapy type (like other SCIG, IVIG, corticosteroids, or plasma exchange) to HyQvia for the maintenance treatment of CIDP, current/future preference for HyQvia, reason for HyQvia or study discontinuation, and details on previous treatment setting/components for other subcutaneous immunoglobulin (SCIG) or intravenous immunoglobulin (IVIG) user only. Users will be presented a maximum of 8 questions at baseline, 2 questions at Month 12, 2 questions if HyQvia is discontinued, and 4 questions if the study is discontinued. The questionnaires will be self-administered.
Treatment Satisfaction With HyQvia as Measured by the Treatment Satisfaction Questionnaire for Medication (TSQM) Short Form-9 | Baseline up to 12 months
  The TSQM is a 9-item questionnaire which assesses domains that include effectiveness, convenience, and global satisfaction. The instrument is self-administered. Response options fall on a 5- or 7-point Likert/Likert-type scale with scores ranging from 0 to 100 and higher scores indicating a higher level of treatment satisfaction.
Health-Related Quality of Life (HRQoL) as Measured by the Chronic Acquired Polyneuropathy Patient Reported Index (CAP-PRI) | Baseline up to 12 months
  The CAP-PRI is a disease-specific HRQoL measure designed to assess diabetic polyneuropathy. This 15-item questionnaire assesses various life domains including physical and social functioning, pain, and emotional well-being. Items will be scored 0 (not at all), 1 (a little bit), or 2 (a lot). Individual scores within the CAP-PRI may be summed to a total score ranging from 0 to 30 that indicates the level of disease impairment, with higher scores representing higher degrees of impairment.
CIDP Signs, Symptoms, and Impacts, as Measured by the Inflammatory Rasch-built Overall Disability Scale (I-RODS) | Baseline up to 12 months (HyQvia or study discontinuation)
  The I-RODS is a linearly weighted scale developed to capture activity and social participation limitations in participants with Guillain-Barré syndrome and CIDP. This 24-item questionnaire assesses domains that include activity and social participation. Response options include a categorical rating scale where 0 is "Not possible to perform," 1 is "Possible with some difficulty," and 2 is "Possible, without any difficulty," with a lower score indicating more severe activity and social participation limitations.
Productivity as Measured by the Work Productivity and Activity Impairment (WPAI) | Baseline up to 12 months
  The WPAI is a 6-item questionnaire that assesses domains that include absenteeism (missing work), presenteeism (impaired productivity at work), overall work performance (combined absenteeism and presenteeism), and non-work activities (activity impairment. Outcomes as measured by the WPAI are expressed as impairment percentages i.e., 0% (best) to 100% (worst), with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes.

SECONDARY OUTCOMES:
Number of Participants With Serious Adverse Events (SAEs) and All Non-serious Adverse Events (AEs) Causally or Temporally Relationship to HyQvia Treatment | Baseline up to 12 months
  SAE is any untoward medical occurrence that at any dose: results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent, significant disability/incapacity, a congenital abnormality/birth defect, an important medical event in opinion of healthcare provider, may jeopardize the participant or may require intervention to prevent one of other outcomes listed in definition above. Non-serious AEs are the AEs that do not meet SAEs definition. Related AE: AE that follows a reasonable temporal sequence from administration of medication, vaccine, or device (including the course after withdrawal of the medication), and for which a causal relationship is at least a reasonable possibility, i.e., relationship cannot be ruled out, although factors other than medication, vaccine or device, such as underlying diseases, complications, concomitant drugs and concurrent treatments, may also have contributed.
Number of Participants With Adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) Increase of >=1 point Relative to the Baseline | Baseline up to 12 months
  The INCAT disability score is a measure of activity limitation. The INCAT disability score ranges from 0 to 10 and is the sum of arm and leg disability each rated between 0 and 5 (where arm = 0 indicates 'no upper limb problems' and arm = 5 indicates 'inability to use either arm for any purposeful movement', and leg = 0 indicates 'walking not affected', and leg = 5 indicates 'restricted to wheelchair, unable to stand and walk a few steps with help'). Thus, a higher INCAT disability score indicates greater disability. The adjusted INCAT disability score remains identical to INCAT disability score, except that the changes in upper limb function from 0 (normal) to 1 (minor symptoms) are excluded.
Change From Baseline in Adjusted INCAT Disability Score | Baseline up to 12 months
  The INCAT disability score is a measure of activity limitation. The INCAT disability score ranges from 0 to 10 and is the sum of arm and leg disability each rated between 0 and 5 (where arm = 0 indicates 'no upper limb problems' and arm = 5 indicates 'inability to use either arm for any purposeful movement', and leg = 0 indicates 'walking not affected', and leg = 5 indicates 'restricted to wheelchair, unable to stand and walk a few steps with help'). Thus, a higher INCAT disability score indicates greater disability. The adjusted INCAT disability score remains identical to INCAT disability score, except that the changes in upper limb function from 0 (normal) to 1 (minor symptoms) are excluded.
Change From Baseline in Hand Grip Strength | Baseline up to 12 months
  Grip strength assessments conducted by prescribing physicians using the Martin Vigorimeter or the Jamar Dynamometer (as available at the site and performed per routine clinical practice).
Change from Baseline in Medical Research Council (MRC) Score | Baseline up to 12 months
  The MRC sum score measures muscle strength from both the left and right sides of the body on a scale of 0 to 5. The total MRC sum score ranges from 0 (paralysis) to 60 (normal strength), where higher score indicates better strength.
Change From Baseline in I-RODS Centile Score | Baseline up to 12 months
  The I-RODS is a linearly weighted scale developed to capture activity and social participation limitations in participants with Guillain-Barré syndrome and CIDP. This 24-item questionnaire assesses domains that include activity and social participation. The instrument is self-administered, takes 5-10 minutes to complete, and the data will be collected electronically. Response options include a categorical rating scale where 0 is "Not possible to perform," 1 is "Possible with some difficulty," and 2 is "Possible, without any difficulty," with a lower score indicating more severe activity and social participation limitations.
Treatment Utilization of HyQvia | Baseline, Month 3, Month 6, Month 9, and Month 12 (as available)
  Data will be reported as average total dose per infusion (mg); proportions of participants with dose as prescribed/planned by physician and with at least one ramp-up infusion; average number of ramp-up doses per participant; average infusion duration (minutes); proportions of participants with treatment intervals at every 2, 3, 4, 5, and 6 weeks; average maximum infusion rate (milliliter/hour[mL/h]); average number of infusion sites per infusion; proportion of participants using 6mm, 8mm, 9mm, 12mm, 14mm, 16mm, and other needle lengths; proportions of participants using 23G, 24G, 25G, 26G, 27G, 28G, 29G, 30G, and other needle gauges; proportions of participants using various infusion pump types; proportions of participants receiving infusions at home, hospital, doctor's office, and other; proportions of participants administering infusions by self, caregiver, or HCP; average adherence; proportion of participants who discontinue HyQvia treatment and their reason of discontinuation.
Healthcare Resource Utilization (HCRU) | Baseline, Month 3, Month 6, Month 9, and Month 12 (as available)
  Data will be reported as number of participants with at least one and average number of emergency room visits; number of participants with at least one and average number of outpatient office visits; number of participants with at least one and average number of hospitalizations; average number of emergency room visits due to severity of AEs within 7 business days of an infusion; average number of outpatient office visits due to severity of AEs within 7 business days of an infusion; average number of hospitalizations due to severity of AEs within 7 business days of an infusion; proportions of participants receiving caregiver or HCP support for infusions.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (15):
- United States (9):
  - Samir Macwan MD Inc, Rancho Mirage, California
  - Neuro/Psych Sleep Clinic, San Francisco, California
  - Yale School Of Medicine, New Haven, Connecticut
  - Nova Clinical Research, LLC, Bradenton, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - HSHS St. Elizabeths Hospital, O'Fallon, Illinois
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Wake Forest University - School of Medicine - Central, Winston-Salem, North Carolina
- Denmark (2):
  - Arhus Universtitetshospital, Aarhus N
  - Rigshospitalet, København Ø
- Germany (4):
  - Immanuel Klinik Rudersdorf, Rüdersdorf, Brandenburg
  - Universitaetsklinikum Giessen und Marburg GmbH Standort Marburg, Marburg, Hesse
  - Katholisches Klinikum Bochum gGmbH, Bochum, North Rhine-Westphalia
  - Judisches Krankenhaus Berlin, Berlin

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/72df72a5325d4de2??page=1&idFilter=TAK-771-5008